CLINICAL TRIAL: NCT00637832
Title: Short Chemo Radiotherapy in Follicular Lymphoma Trial of 90Y Ibritumomab Tiuxetan (ZevalinTM) as Therapy for First and Second Relapse in Follicular Lymphoma
Brief Title: Rituximab, Combination Chemotherapy, and Yttrium Y 90 Ibritumomab Tiuxetan in Treating Patients With Relapsed Follicular Non-Hodgkin Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: no information
Sponsor: University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000588042; USCTU-SCHRIFT-06-DOG05-44 (Other: USCTU); USCTU-RHM-CAN0542 (Other: USCTU-RHM); 2007-000222-51 (EudraCT Number); EU-20819 (Other: EU)
Record Dates: First submitted 2008-03-14; First posted 2008-03-18 (Estimated); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Lymphoma
Keywords: recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Prednisolone; Vincristine; ibritumomab tiuxetan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single group (Experimental)
  Interventions: Biological: rituximab; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: prednisolone; Drug: vincristine sulfate; Radiation: yttrium Y 90 ibritumomab tiuxetan

INTERVENTIONS:
Biological: rituximab
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: prednisolone
Drug: vincristine sulfate
Radiation: yttrium Y 90 ibritumomab tiuxetan

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Radiolabeled monoclonal antibodies, such as yttrium Y 90 ibritumomab tiuxetan, can find cancer cells and carry cancer-killing substances to them without harming normal cells. Giving rituximab together with combination chemotherapy and yttrium Y 90 ibritumomab tiuxetan may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving rituximab together with combination chemotherapy and yttrium Y 90 ibritumomab tiuxetan works in treating patients with relapsed follicular non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the response rates in patients with relapsed follicular non-Hodgkin lymphoma treated with short-duration rituximab and combination chemotherapy (R-chemo) followed by rituximab and yttrium Y 90 ibritumomab tiuxetan.

Secondary

* To evaluate the duration of response in patients treated with this regimen.
* To evaluate the quality of response in order to determine the conversion rate from partial response to complete response in patients treated with this regimen.
* To evaluate the toxicity of yttrium Y 90 ibritumomab tiuxetan when administered after 3 courses of R-chemo.

OUTLINE: This is a multicenter study.

* Chemoimmunotherapy (R-CHOP or R-CVP): Patients receive R-CHOP comprising rituximab IV, cyclophosphamide IV, doxorubicin hydrochloride IV, and vincristine IV on day 1 and oral prednisolone on days 1-5. Alternatively, patients who have already been exposed to prior tolerance doses of anthracyclines receive R-CVP comprising rituximab IV, cyclophosphamide IV, and vincristine IV on day 1 and oral prednisolone on days 1-5. Treatment repeats every 3 weeks for up to 3 courses.

Patients with objective evidence of response on CT scan or those with < 25% bone marrow involvement and no signs of bone marrow hypocellularity (< 15%) on bone marrow biopsy proceed to radioimmunotherapy.

* Radioimmunotherapy: Four to 6 weeks after completion of R-CHOP or R-CVP, patients receive rituximab IV followed no more than 4 hours later by yttrium Y 90 ibritumomab tiuxetan IV over 10 minutes.

After completion of study therapy, patients are followed periodically for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed grade 1, 2, or 3 follicular non-Hodgkin lymphoma

  * Stage II, III, or IV disease (according to the Ann Arbor staging system)
* CD20-positive disease
* Initial disease bulk ≤ 10 cm
* In first or second relapse after prior treatment with a rituximab-containing chemotherapy regimen (R-chemo) or chemotherapy alone

  * Relapse must have occurred ≥ 6 months after completion of R-chemo

    * Relapse that occurred < 6 months after completion of chemotherapy alone allowed
* Has at least one of the following symptoms requiring initiation of treatment:

  * Nodal mass > 5 cm in its greater diameter
  * B symptoms
  * Elevated serum lactate dehydrogenase (LDH) or β2-microglobulin
  * Involvement of ≥ 3 nodal sites (each with a diameter > 3 cm)
  * Symptomatic splenic enlargement
  * Compressive syndrome
* No primary refractory disease
* No large pleural or peritoneal effusions
* No CNS disease

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 6 months
* Absolute granulocyte count ≥ 1,500/mm³
* Platelet count ≥ 1,000/mm³
* Serum creatinine < 1.5 times upper limit of normal (ULN)
* Total bilirubin < 1.5 times ULN
* AST < 5 times ULN
* No active obstructive hydronephrosis
* No evidence of active infection requiring IV antibiotics
* No advanced heart disease or other serious illness that would preclude study evaluation
* No known HIV infection
* No human anti-mouse antibody (HAMA) reactivity
* No known hypersensitivity to murine antibodies or proteins
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 12 months after completion of study treatment
* No other prior malignancy, except for adequately treated skin cancer, cervical cancer in situ, or other cancer for which the patient has been disease-free for 5 years

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 4 weeks since prior investigational drugs and recovered
* No prior radioimmunotherapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-04-01 (Actual); Primary Completion 2015-01-06 (Actual); Study Completion 2015-01-06 (Actual)

PRIMARY OUTCOMES:
Overall response rate, including combined complete response and partial response

SECONDARY OUTCOMES:
Time to disease progression
Time to next treatment
Response duration in patients with responding disease
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Tim Illidge, Principal Investigator — The Christie NHS Foundation Trust
Locations (5):
- United Kingdom (5):
  - Christie Hospital, Manchester, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Dorset Cancer Centre, Poole Dorset, England
  - Southampton General Hospital, Southampton, England
  - Saint Bartholomew's Hospital, London

REFERENCES:
- [Derived] Illidge TM, McKenzie HS, Mayes S, Bates A, Davies AJ, Pettengell R, Stanton L, Cozens K, Hampson G, Dive C, Zivanovic M, Tipping J, Gallop-Evans E, Radford JA, Johnson PW. Short duration immunochemotherapy followed by radioimmunotherapy consolidation is effective and well tolerated in relapsed follicular lymphoma: 5-year results from a UK National Cancer Research Institute Lymphoma Group study. Br J Haematol. 2016 Apr;173(2):274-82. doi: 10.1111/bjh.13954. Epub 2016 Feb 5. PMID 26849853